CLINICAL TRIAL: NCT04154566
Title: Influence of Aerobic Exercise on Inhibitory Control of Excutive Function in Spastic Hemiplegic Cerebral Palsy: A Randomized Controlled Trail
Brief Title: Influence of Aerobic Exercise on Inhibitory Control of Excutive Function in Spastic Hemiplegic C.P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohammed E. Ali, Ph. D Candidate., Lecturer, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P. T. REC/012/002278
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Spastic Hemiplegic Cerebral Palsy
Keywords: Hemiplegic cerebral palsy; inhibitory control of executive functions.; aerobic exercise.
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: They were assigned randomly into two equal groups. Group (A) the study group received aerobic exercise in addition to selected physical therapy program. And group (B) the control group received the same selected physical therapy program only. The treatment was conducted for one hour, three times / weak for three successful months.
Who Masked: Outcomes Assessor
Masking Description: Blinding process to participants and care providers was impossible due to the nature of intervention therapy. Data were analyzed by an impartial statistician (outcomes assessor), referring to each arm with an encoded name: Group A (control group) and Group B (study group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the study group (Experimental): Group (A) the study group received aerobic exercise in addition to selected physical therapy program which contain strengthening exercises for upper limb and lower limb muscles, stretching exercises for elbow extensors, hand supinator, wrist extensors, knee extensors and ankle dorsiflexors, balancing exercises, coordination exercises and gait training exercises in open environment.
  Interventions: Other: Aerobic Exercises
- the control group (No Intervention): group (B) the control group received the same selected physical therapy program which contain strengthening exercises for upper limb and lower limb muscles, stretching exercises for elbow extensors, hand supinator, wrist extensors, knee extensors and ankle dorsiflexors, balancing exercises, coordination exercises and gait training exercises in open environment only.

INTERVENTIONS:
Other: Aerobic Exercises — Aerobic exercise refers to exercise that involves or improves oxygen consumption by the body. It is the type of activity that uses large muscle groups. Its performance is in a continuous and rhythmic way with a main goal to make the heart and lungs work harder than they do when the person at rest
  Arms: the study group

SUMMARY:
The study was conducted to assess the influence of aerobic exercise on inhibitory control of executive functions in spastic hemiplegic cerebral palsy.

DETAILED DESCRIPTION:
Inhibitory control of executive functions (EF) is one of the main specific cognitive impairments that affect children with cerebral palsy, cognitive skills begin to develop in infancy and continuing through the pre-school years, childhood and into adolescence it changes across the lifespan of an individual and has great effect on their participation and quality of life. The aim of study was to assess the influence of aerobic exercise on inhibitory control of executive functions in spastic hemiplegic cerebral palsy. Sixty children with spastic hemiplegic cerebral palsy were enrolled in this study and were assessed for eligibility. Their aged ranged from seven and eleven years. They were assigned randomly into two equal groups. Group (A) the study group received aerobic exercise in addition to selected physical therapy program. And group (B) the control group received the same selected physical therapy program only. The treatment was conducted for one hour, three times / weak for three successful months. Eriksen flanker test and Stroop Color-Word test were used to assess inhibitory control of EF pre and post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Their aged ranged from seven and eleven years.
* they were from both sexes.
* they have left side hemiplegic cerebral palsy.
* they were able to walk independently.

Exclusion Criteria:

* children with visual or auditory problems.
* children with history of drug intake that may affect the cognitive function.
* medically unstable children especially with cardiovascular disorders.
* uncooperative children.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
The mean values of the Flanker test accuracy, congrunent reaction time and incongruent reaction time | Eriksen flanker test was assessed at day 0, 90.
  the Eriksen flanker task is a set of response inhibition tests used to assess the ability to suppress responses that are inappropriate in a particular context. The target is flanked by non-target stimuli which correspond either to the same directional response as the target (congruent flankers), to the opposite response (incongruent flankers), or to neither (neutral flankers).
The mean values of the Stroop test accuracy, congrunent reaction time and incongruent reaction time | Stroop Color-Word test was assessed at day 0, 90.
  The Stroop Color and Word Test (SCWT) is a neuropsychological test extensively used to assess the ability to inhibit cognitive interference that occurs when the processing of a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute, well-known as the Stroop Effect.

CONTACTS AND LOCATIONS:
Overall Officials: Nehad A. Abo-zaid, PhD, Principal Investigator — South Valley University, Faculty of Physical Therapy; Mohammed E. Ali, PhD student, Principal Investigator — South Valley University, Faculty of Physical Therapy
Locations (1):
- South Valley University, Faculty of Physical Therapy, Qina, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sutoo D, Akiyama K. Regulation of brain function by exercise. Neurobiol Dis. 2003 Jun;13(1):1-14. doi: 10.1016/s0969-9961(03)00030-5. PMID 12758062
- [Background] Chang YK, Labban JD, Gapin JI, Etnier JL. The effects of acute exercise on cognitive performance: a meta-analysis. Brain Res. 2012 May 9;1453:87-101. doi: 10.1016/j.brainres.2012.02.068. Epub 2012 Mar 4. PMID 22480735
- [Background] Wecker NS, Kramer JH, Wisniewski A, Delis DC, Kaplan E. Age effects on executive ability. Neuropsychology. 2000 Jul;14(3):409-14. doi: 10.1037//0894-4105.14.3.409. PMID 10928744
- [Background] Kluding PM, Tseng BY, Billinger SA. Exercise and executive function in individuals with chronic stroke: a pilot study. J Neurol Phys Ther. 2011 Mar;35(1):11-7. doi: 10.1097/NPT.0b013e318208ee6c. PMID 21475079
- [Result] Rosenbaum P, Paneth N, Leviton A, Goldstein M, Bax M, Damiano D, Dan B, Jacobsson B. A report: the definition and classification of cerebral palsy April 2006. Dev Med Child Neurol Suppl. 2007 Feb;109:8-14. PMID 17370477
- [Result] Garne E, Dolk H, Krageloh-Mann I, Holst Ravn S, Cans C; SCPE Collaborative Group. Cerebral palsy and congenital malformations. Eur J Paediatr Neurol. 2008 Mar;12(2):82-8. doi: 10.1016/j.ejpn.2007.07.001. Epub 2007 Sep 19. PMID 17881257
- [Result] Holmefur M, Kits A, Bergstrom J, Krumlinde-Sundholm L, Flodmark O, Forssberg H, Eliasson AC. Neuroradiology can predict the development of hand function in children with unilateral cerebral palsy. Neurorehabil Neural Repair. 2013 Jan;27(1):72-8. doi: 10.1177/1545968312446950. Epub 2012 Jun 6. PMID 22677505
- [Result] Arner M, Eliasson AC, Nicklasson S, Sommerstein K, Hagglund G. Hand function in cerebral palsy. Report of 367 children in a population-based longitudinal health care program. J Hand Surg Am. 2008 Oct;33(8):1337-47. doi: 10.1016/j.jhsa.2008.02.032. PMID 18929198
- [Result] Hielkema T, Hadders-Algra M. Motor and cognitive outcome after specific early lesions of the brain - a systematic review. Dev Med Child Neurol. 2016 Mar;58 Suppl 4:46-52. doi: 10.1111/dmcn.13047. PMID 27027607
- [Result] McClelland MM, Cameron CE, Duncan R, Bowles RP, Acock AC, Miao A, Pratt ME. Predictors of early growth in academic achievement: the head-toes-knees-shoulders task. Front Psychol. 2014 Jun 17;5:599. doi: 10.3389/fpsyg.2014.00599. eCollection 2014. PMID 25071619
- [Result] Wolf SA, Kronenberg G, Lehmann K, Blankenship A, Overall R, Staufenbiel M, Kempermann G. Cognitive and physical activity differently modulate disease progression in the amyloid precursor protein (APP)-23 model of Alzheimer's disease. Biol Psychiatry. 2006 Dec 15;60(12):1314-23. doi: 10.1016/j.biopsych.2006.04.004. Epub 2006 Jun 27. PMID 16806094
- [Result] Pereira AC, Huddleston DE, Brickman AM, Sosunov AA, Hen R, McKhann GM, Sloan R, Gage FH, Brown TR, Small SA. An in vivo correlate of exercise-induced neurogenesis in the adult dentate gyrus. Proc Natl Acad Sci U S A. 2007 Mar 27;104(13):5638-43. doi: 10.1073/pnas.0611721104. Epub 2007 Mar 20. PMID 17374720
- [Result] McMorris T, Hale BJ. Differential effects of differing intensities of acute exercise on speed and accuracy of cognition: a meta-analytical investigation. Brain Cogn. 2012 Dec;80(3):338-51. doi: 10.1016/j.bandc.2012.09.001. Epub 2012 Oct 11. PMID 23064033
- [Result] Gellish RL, Goslin BR, Olson RE, McDonald A, Russi GD, Moudgil VK. Longitudinal modeling of the relationship between age and maximal heart rate. Med Sci Sports Exerc. 2007 May;39(5):822-9. doi: 10.1097/mss.0b013e31803349c6. PMID 17468581
- [Result] Boyd RN, Davies PS, Ziviani J, Trost S, Barber L, Ware R, Rose S, Whittingham K, Sakzewski L, Bell K, Carty C, Obst S, Benfer K, Reedman S, Edwards P, Kentish M, Copeland L, Weir K, Davenport C, Brooks D, Coulthard A, Pelekanos R, Guzzetta A, Fiori S, Wynter M, Finn C, Burgess A, Morris K, Walsh J, Lloyd O, Whitty JA, Scuffham PA. PREDICT-CP: study protocol of implementation of comprehensive surveillance to predict outcomes for school-aged children with cerebral palsy. BMJ Open. 2017 Jul 12;7(7):e014950. doi: 10.1136/bmjopen-2016-014950. PMID 28706091

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-27): https://cdn.clinicaltrials.gov/large-docs/66/NCT04154566/Prot_SAP_001.pdf